CLINICAL TRIAL: NCT05008770
Title: Trial in Elderly With Musculoskeletal Problems Due to Underlying Sarcopenia - Faeces to Unravel Gut and Inflammation Translationally
Acronym: TEMPUS-FUGIT
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Research Foundation Flanders (Other); KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s65127; B32220221000449 (Registry Identifier: Belg. Regnr.)
Record Dates: First submitted 2021-07-28; First posted 2021-08-17 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Sarcopenia
Keywords: gut microbiota; gut-muscle axis; healthy ageing; intestinal inflammation; systemic inflammation; gut microbiome
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Stool, blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults without sarcopenia: Healthy volunteers aged 65+ years who do not fulfill diagnostic criteria for sarcopenia, according to the revised European Working Group on Sarcopenia in Older People (EWGSOP2)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The overall aim of the TEMPUS-FUGIT study is to assess gut microbiota composition in older persons without sarcopenia and to determine the relationship with and between intestinal and systemic inflammation and with sarcopenia-defining parameters (muscle mass, muscle strength and physical performance). The gut microbiota of older persons without sarcopenia (included in TEMPUS-FUGIT) will be compared with the gut microbiota of older people with sarcopenia, participating in the Exercise and Nutrition for Healthy AgeiNg (ENHANce) study (NCT03649698).

ELIGIBILITY:
Inclusion Criteria:

* Male or female persons without probable, confirmed or severe sarcopenia according to the European Working Group on Sarcopenia in Older People (EWGSOP2): no reduced muscle strength measured by chair stand test or hand grips strength
* 65 years or older
* Community-dwelling elderly or assisted living
* Dutch speaking

Exclusion Criteria:

* Impairments/diseases that affect performance of daily activities
* Persons who are systematically physically active (e.g. routine or organized sports activities) or who followed a physical activity training program (e.g., rehabilitation program) in the last 6 months (systematically = twice or more/week)
* Diagnosis of diabetes mellitus, measured by fasting glucose ≥126 mg/dL or HbA1C ≥ 6.5% at screening or in recent (maximum 3 months old) lab report
* Use of antibiotics in the last 3 months
* Gastrointestinal cancer (active or treated in the last 5 years)
* No freezer at home available

After the screening visit, included persons will be invited for a test visit.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Study Population: Healthy volunteers (aged 65+ years) without probable, confirmed or severe sarcopenia (according to the EWGSOP2), matched according to gender, age and BMI with participants of ENHANce (NCT03649698)
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota composition | Baseline
  Gut microbiota composition (measured through 16S ribosomal RNA (rRNA) gene sequencing).
Intestinal inflammation | Baseline
  Markers of intestinal inflammation: fecal calprotectin, lactoferrin, S100A12
Systemic inflammation | Baseline
  Markers of inflammation in blood samples: C reactive protein (hs-CRP), sedimentation rate, Interleukin 6 (IL-6), IL-4, IL-13, IL-1b, Tumor necrosis factor alpha

SECONDARY OUTCOMES:
Physical performance | Baseline
  Short Physical Performance Battery (SPPB) score
Physical performance (gait speed) | Baseline
  gait speed (expressed in m/s)
Muscle strength (upper limbs) | Screening; baseline
  Handgrip strength measured with Jamar dynamometer (expressed in kg)
Muscle strength (lower limbs) | Screening; baseline
  Chair stand test
Muscle mass (BIA) | Baseline
  Appendicular lean mass measured with a Dual-energy X-ray absorptiometry (DXA) scan
Muscle mass (DXA) | Baseline
  Appendicular lean mass measured with bioelectrical impedance analysis
Dietary intake | Baseline
  Food diaries will help to evaluate dietary protein and fatty acids intake
Urinary nitrogen | Baseline
  Urinary nitrogen
Functional status | Baseline
  Frailty scale according to Fried et al. (2001)
Functional status (ADL) | Baseline
  Activities of daily living (Barthel index)
Balance | Baseline
  Mini-Balance Evaluation Systems Test (Mini-BESTest)
Physical activity | Baseline
  Time of physical activity throughout the day measured with MoveMonitor+
Health-related quality of life (SF-36) | Baseline
  Measured trough the Short Form Health Questionnaire (SF-36) Quality of Life)
Health-related quality of life (SarQoL) | Baseline
  SarQoL(Sarcopenia Quality of Life)
Cognitive status (MMSE) | Baseline
  Mini-Mental State Exam (MMSE)
Cognitive status (RBANS) | Baseline
  Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)

CONTACTS AND LOCATIONS:
Overall Officials: Evelien Gielen, PhD MD, Principal Investigator — Gerontology and Geriatrics, Department of Public Health and Primary Care, KULeuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lapauw L, Dupont J, Amini N, Vercauteren L, Verschueren S, Tournoy J, Raes J, Gielen E. Trial in Elderly with Musculoskeletal Problems due to Underlying Sarcopenia-Faeces to Unravel the Gut and Inflammation Translationally (TEMPUS-FUGIT): protocol of a cross-sequential study to explore the gut-muscle axis in the development and treatment of sarcopenia in community-dwelling older adults. BMC Geriatr. 2023 Sep 26;23(1):599. doi: 10.1186/s12877-023-04291-5. PMID 37752426